CLINICAL TRIAL: NCT05491863
Title: Effects of Trunk Stability Exercises on Hand Function in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0710
Record Dates: First submitted 2022-07-24; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Palsy
Keywords: trunk stability; hand function
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: . Participants were randomly assigned to the experimental group or control group after a baseline assessment with a lottery ticket and an opaque envelope containing the same number of folded papers labeled "control" or "intervention." Each participant took a piece of paper that identified their group and gave it to the researchers without seeing what was written. Participants were not notified which group was assigned to
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers who evaluated the participants were not informed of how the participants were grouped. Participants were informed that they would receive one of two different interventions without indicating which group should undergo trunk stability or conventional physiotherapy program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conservative physiotherapy plan (Active Comparator): Postural and Proprioceptive facilitation,walking ,jumping and staircase activity
  Interventions: Other: conservative physiotherapy plan; Other: trunk stability exercise plan
- Trunk stability exercise plan (Experimental): Trunk stability exercises including proprioception,balance and stability.
  Interventions: Other: conservative physiotherapy plan; Other: trunk stability exercise plan

INTERVENTIONS:
Other: conservative physiotherapy plan — Physiotherapy plan consist of following exercises, Postural and Proprioceptive facilitation like weight-bearing actions for the upper and lower extremities. Sit to stand, standing , holding on to stand, free arms standing up, holding on standing and asked the patient to lift one leg, one leg standing, standing on balance board,Straight and sideways parallel bar walk, For the effected body side jumping on stable and dynamic surface,Upstairs and down stair activity performed on staircase.This program was given for 40 minutes with a rest period of 2 minutes between each group of exercises, 4 days a week for 8 weeks (32 sessions)
Other: trunk stability exercise plan — trunk stability exercise plan consist of three levels, Proprioception included supine abdominal draw was performed in 1st simple level ,3 sets per 20 repetitions were performed, A double knee to chest abdominal draw was performed with 3 sets per 20 repetition, Supine twist with 3 sets per 20 repetitions was performed.Balance training included pelvic bridging was 2nd complicated level performed with 3 sets per 4-6 repetitions,Twists with a medicine ball were performed with 3 sets per 10-20 repetitions.
  for Stability Bridging with head lied on physio ball was performed in 3rd difficult level when holding the position for 4 to 6 seconds, then relaxed slowly for same time with 3 sets per 10 to 20 repetitions, Prone bridging was performed with 3 sets per 4 to 6 repetitions.
  There was a 30 seconds to 1 minute break between the sets.This program was given for 1 hour with a rest period of 2 minutes between each group of exercises, 4 days a week for 8 weeks (32 sessions)

SUMMARY:
Rationale of this research is to evaluate the outcome of trunk stabilizing exercises on the fine motor skills of subjects with hemiplegic CP. The significance of this study is to identify how much core stability exercises improve hand function. This study will help gather evidence on the practice of core stabilizing exercises to improve hand function so that it can help both physicians and patients.

DETAILED DESCRIPTION:
Cerebral palsy is a permanent damage in early brain in fetus which leads to movement disorder. The most frequent reason of bodily incapacity is cerebral palsy in pediatric population. CP children have difficulty maintaining dynamic and static trunk stability, which leads to affect sitting, standing, reaching and walking. Hemiplegic Cerebral palsy patients are challenged by fine motor skills, like gripping or object handling, which are essential for activities of daily life.the purpose of the study was to evaluate the effects of trunk stability exercises on hand function in children with cerebral palsy.It was a randomized, controlled trial, conducted among hemiplegic cerebral palsy patients. Sample size was 26 by using Epitool software. Participants were randomly assigned to the intervention or control group after a baseline assessment with a lottery ticket and an opaque envelope. All participants in both groups were evaluated on three occasions: (i) baseline (ii) post-intervention and (iii) after 4 weeks follow to assess long term effects.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female were included
* Age group 6 to 18 years.
* Medical diagnosis of hemiplegic cerebral palsy assured.
* Unilateral Movement deficit (less than 2.5) on amount of use scale on MAL (motor activity log).
* Level 1 to 3 on manual ability classification system (MACS).
* Mild to moderate spasticity of upper extremity (MAS grade 1 to 2.)
* GMCS level I-II.
* Subjects were cognitively capable and competent to follow the instructions

Exclusion Criteria:

* Patients with altered conscious level.
* Previous surgery or pain in upper limbs.
* Rigid contracture and fixed deformities in the spine
* Auditory / vision problem.
* Previous Botulinum Toxin-A injections in upper limb.
* Cardio-respiratory problem

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Trunk Control Meaurment Scale | 12 week
  The trunk control measurement scale measures two mechanism of trunk control throughout functional activities. First level begins with smooth base of support and it ends on dynamic service to assess balance of body.15 items performed with the sub scales that consist of 5, 7 and 3 activities respectively. Total score ranges from 0 to 58 on scale.
ABILHAND-kids (Manual Ability Measure) | 12 week
  ABILHAND-Kids questionnaire is valuable tool to assess a child's unimanual and bimanual upper limb activities. This 21 items hand use scale with total 63 score prestents low to high performance of fine motor .
CHEQ (Children's hand-use experience's questionnaire) | 12 weeks
  Children's Hand-use Experience Questionnaire has been developed to capture kid's perceived quality of performance when using the affected hand in these situations. CHEQ is an internet based questionnaire containing 29 items with (bimanual activities) presented one by one in random order .score ranges from 0 to 100 representing better function with higher score .

SECONDARY OUTCOMES:
UE MAL | 12 weeks
  It consists of both the AS and HW scales are used during all test administrations, except for the periodic administrations of MAL during treatment, when only the HW scale is used. In all administrations except those done during treatment, begin with AS scale and ask participants to rate all task using the AS scale first the participant than rates all tasks perform with the HW scale
Manual ability classification system | 12 weeks
  It's a 5 level ordinal classification system which describes the manual ability of children aged 4 to 18 years with cerebral palsy. When children holds objects in typical activities, MACS levels describe the collaborative use of both hands together in daily life activities .As a classification system the purpose of MACS is to discriminate meaningfully on child's manual ability to handle objects in daily living. It's not an outcome measure or diagnostic tool
Modified ash worth scale (MAS) | 12 weeks
  The original ash worth scale by Bryan Ashworth was a five point numerical scale that graded spasticity from 0 to 4, with zero being no resistance and 4 being a limb rigid in flexion or extension. In 1987 when while performing a study to exam reliability of manual tests of elbow flexor muscle spasticity, Bohannon and Smith modified the ash worth scale by adding 1+ to scale to increase sensitivity. Since modified ash worth scale has been applied in clinical practice and research as measure/grade muscle spasticity

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Shafique, tDPT, Principal Investigator — Riphah International University
Locations (1):
- Rising sun institute for special children, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No